CLINICAL TRIAL: NCT04297449
Title: Prospective 2-year Data Collection of the First 10 Patients After Ankle Spacer
Brief Title: Prospective 2-year Data Collection of the First 10 Patients After Ankle Spacer Implantation
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 8198_MPG_23b_2018
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Osteochondritis Dissecans
Keywords: Osteochondral defects (OCD) of the talus; Ankle Spacer; osteoarthritis of the ankle joint
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteochondral defects (OCD) of the talus are pathologic lesions of the talar cartilage and its subchondral bone and might severely deteriorate the quality of life. For the treatment of multiple and/or large talar OCDs and in patients with failed previous surgical treatment the Ankle Spacer was developed. Six patients are included in a prospective clinical and radiological study with a follow-up of two years.

DETAILED DESCRIPTION:
One surgeon in the investigator's center implanted 10 Ankle Spacers between April 2018 and October 2020. The average age was 41.7 years (20 - 70 years). All patients get a standard followed-up at 6 weeks, 12 weeks. After the first four patients, all following patients are enrolled in a prospective study and where followed up after 1 and 2 years additionally. The American Orthopaedic Foot and Ankle Society (AOFAS) Score, the Foot and Ankle Outcome Score (FAOS), the European Foot and Ankle Score (EFAS), the Visual Analogue Scale (VAS) for pain are collected. Radiographic parameters such as implant loosening, cystic changes, lateral/medial prominence of the implant, congruency to the talar rounding, progression of osteoarthritis or bone ware of the tibia plafond are recorded. The Ankle Spacer is a one-piece implant system that replaces the articulating upper talus surface of the tibio-talar joint, and offers several implant sizes in order to fit to the different talus sizes. It is anatomically designed to the native upper talus surface to provide an optimal fit to the distal articular surface. It has a rough titanium plasma spray (TPS) coated under surface with two posts and spikes for implant fixation. The rough surface enables secondary fixation by means of bone ingrowth and the spikes at the posterior part of the prosthesis allowing for optimal adherence of the implant and for minimal iatrogenic damage upon fixation. By these means, the anatomical situation and the natural congruency of the ankle joint are mirrored to an optimal extent.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18-80 years
* Indication for implantation of the ankle spacer

Exclusion Criteria:

* Florid infections
* Relevant circulatory disorders on the affected leg
* Malposition of the OSG (upper ankle Joint) greater than 5 ° varus or valgus
* Fractures of the OSG or near the ankle that were less than 6 months ago
* Obesity with a BMI greater than 30 kg / m2
* Known insulin-dependent diabetes mellitus
* Known rheumatoid Arthritis
* Osteoarthritis of the OSG II ° or higher according to Kellgren / Lawrence
* Deformation of the OSG, which does not allow implantation of the ankle spacer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The average age is 41.7 years (20 - 70 years). Patients with multiple and/or large talar osteochondral defects (OCD) and patients with failed previous surgical treatment for OCD or osteoarthritis of the talus with up to grade two (Kellgren-Lawrence-Score) osteoarthritis on the tibial site are included.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Prospective 2-year Data Collection of the First 10 Patients after Ankle Spacer Implantation | 2 Years
  Prospective 2-year Data Collection of the First 10 Patients after Ankle Spacer Implantation

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Lerch, PD Dr., Principal Investigator — Orthopädische Klinik der Medizinischen Hochschule Hannover im DIAKOVERE Annastift
Locations (1):
- Orthopädische Klinik der Medizinischen Hochschule Hannover im DIAKOVERE Annastift, Hanover, Lower Saxony, Germany